CLINICAL TRIAL: NCT03427021
Title: A Randomized Study to Establish the Efficacy of Oral Ice Exposure During Oxaliplatin Infusion in Preventing Oral Cold Sensitivity
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: final study report has been completed and submitted
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 28216
Record Dates: First submitted 2018-01-30; First posted 2018-02-09 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: GI Patients on Oxaliplatin Containing Regimen
MeSH Terms: interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): will be treated with consistent exposure to oral ice
  Interventions: Drug: Oxaliplatin
- Arm B (Active Comparator): Will not be treated with consistent exposure to oral ice.
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — Infusion

SUMMARY:
The main purpose of this study is to evaluate whether exposure to ice chips in the mouth (oral ice chips) during oxaliplatin treatment prevents or reduces symptoms of cold sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥18 years of age will be enrolled.
* Patients must have histologic confirmation of a solid tumor malignancy that will be treated with a regimen that contains full-dose oxaliplatin.
* Patients may be receiving treatment in the neoadjuvant, adjuvant or metastatic setting.
* Patients must be treatment-naïve to platinum-agents at the time of enrollment. Prior treatment with non-platinum agents is permitted.

Exclusion Criteria:

* Any active intraoral infection, including yeast infection (thrush) or active oral herpes simplex virus at the time of enrollment.
* Patients may not have dentures.
* Patients may not have a disorder that may result in altered taste sensation at baseline. This includes but is not limited to: persistent dry mouth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
overall intraoral cold sensitivity score | a minimum of four cycles (2 months) and a maximum of 12 cycles (6 months)
  graded 0 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Kim Reiss Binder, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States